CLINICAL TRIAL: NCT03111771
Title: Mitochondrial Activity and Myosteatosis in the Cachexia of Cancers of the Upper Aerodigestive Tract
Acronym: MYOMEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-313; 2016-A00611-50 (Other: 2016-A00611-50)
Record Dates: First submitted 2017-03-31; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cancer of Upper Aerodigestive Pathways; Cachexia
Keywords: Cancer; Cachexia; Myosteatosis; Mitochondrial activity; Upper aerodigestive pathways; Lipotoxicity
MeSH Terms: conditions — Cachexia; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group K +: Group K +: cancer of the upper aerodigestive tract with or without cachexia
  Interventions: Procedure: carcinological surgery
- Group K-: Group K-: absence of cancer and absence of cachexia
  Interventions: Procedure: cervical surgery
- Control group: The MYOMEC study includes the inclusion of healthy patients (to form a control group
  Interventions: Procedure: carcinological surgery; Procedure: cervical surgery

INTERVENTIONS:
Procedure: carcinological surgery — carcinological surgery for Group K +
  Groups: Control group; Group K +
Procedure: cervical surgery — cervical surgery for Group K-
  Groups: Control group; Group K-

SUMMARY:
Loss of muscle mass (scientific term: cachexia) affects about 80% of patients with advanced cancer and impacts their prognosis by decreasing tolerance and response to treatment, decreasing quality of life and survival. The prognosis in these patients depends directly on the importance of the loss of muscle mass. Preserving it is therefore an essential therapeutic objective. It is therefore important to understand perfectly the mechanism of this muscular loss. The accumulation of fat in the muscle (scientific term: myosteatosis) could be a mechanism responsible for this loss of muscle mass. It is indeed a hypothesis proved on animal models. Moreover, it has recently been shown that more the cancer patient loses weight, more his muscle contains fat. This lets think that this deposit of fat in the muscle would be directly related to the loss of muscle mass. All of these observations could not be clearly established in humans and investigators are seeking by this study to illuminate these mechanisms at the human level. A better understanding of these mechanisms would allow investigator to set up targeted treatments against the accumulation of fat in the muscle, which would significantly improve the quality of life of patients with cancer of the aerodigestive pathways and their chances of recovery.

The MYOMEC study includes the inclusion of healthy patients (to form a control group) but also patients with cancer of the upper aero-digestive tract. The study will be divided into two parts: clinical examination and nutritional evaluation the day before surgery at the time of the participants' admission to hospital and then the biological samples during surgery. The nutritional examination consists in collecting the morphological data of the patient, namely:

Its weight, size, calculation of the body mass index Tests of muscular strength (wearing weight of 1, 2 and 3 kilos) Measurement of the percentage of fat mass and lean mass (Impedancemetry)

In this study, participants benefit from the following investigations:

* Clinical examination complete with elaboration of the clinical nutritional status, realized the day before the surgical intervention in hospitalization.
* Elaboration of the radiological nutritional status by a complementary analysis of the scanner envisaged in the balance of extension of the disease
* Performing surgical site sampling during surgery without additional invasive procedure and under general anesthesia. It will be realized:

A muscle biopsy of the sterno-cleido-mastoid muscle (neck muscle) (maximum volume 5 mm3), A tumor biopsy (maximum volume 5mm3). A blood sample (maximum volume 5ml)

No invasive procedure, supplemental examination or additional consultation is required for the whole off-set study for the extensive muscular percutaneous biopsy regarding which additional patient agreement will be required. No additional follow-up is required when participating in this study. Participation in this study does not entail any particular constraint or additional treatment. The duration of the patient's participation is defined as follows: from the date of the preoperative consultation or from the consultation of announcement until his / her discharge from hospital. The exclusion period defined in this study extends from the date of inclusion of the patient to the date of the surgical procedure, during which time the patient can not participate in another clinical research protocol.

DETAILED DESCRIPTION:
Malnutrition is characterized by a negative energy balance due to a deep skeletal muscular loss, which is itself secondary to the reduction of intake and metabolic abnormalities aggravating the loss of weight. Sarcopenia is defined as the loss of muscle mass, the consequences of which are a decrease in muscle strength and physical performance .Cachexia, identified in many chronic diseases (renal insufficiency, heart failure, diabetes, COPD), is the result of an imbalance between proteolysis and proteogenesis and can be defined as a multifactorial syndrome characterized by a weight loss resulting mainly from a loss of lean mass, in particular muscle mass, which is not reversible by an adequate nutritional contribution and which leads to functional abnormalities.

Cancers of the ENT sphere represent about 15% of all cancers in men and 2% in women. They mainly concern subjects between 45 and 70 years of age with a predominant role of ethylo-tobacco poisoning. Patients with upper aero-digestive tract cancers are particularly prone to malnutrition on the part of the tumor itself but also on the context (ethylo-tobacco intoxication, sedentary behavior, poor general condition), tumor localization involving reduction of intake (Mechanical obstruction, anorexia, pain), but also after treatment (chemotherapy, radiotherapy, surgery).

Cancer cachexia affects approximately 80% of patients with advanced cancer and impacts their prognosis by increasing morbidity and mortality, decreased tolerance and response to treatment , decreased quality of life and decreased survival. Its prognosis depends on the extent of the loss of muscle mass. It is generally reported for a patient with a weight loss superior than 5% of its initial weight over the last 6 months, with 3 stages described: Pre-cachexia stage, clean cachexia stage, refractory cachexia stage. It is characterized, among other things, by the development of systemic inflammation and tumor cell lines and tumor cells from cancer patients have been shown to produce pro-inflammatory cytokines ( IL-6, IL-8).

The loss of skeletal muscle mass, up to 75% in severe malnutrition is related to an acceleration of muscle catabolism and an alteration of muscle protein anabolism, mediated by large tumor signals and leads to a decrease in performans status, decrease in overall survival, increase in susceptibility to toxicity of chemotherapy, and increase in exposure to long-term hospital stays.

This muscular loss is the result of an increase in proteolysis phenomen but also of a decrease in protein synthesis. The main proteolytic pathways are the calpain-calcium-dependent pathway, the lysosomal pathway and the ubiquitin-proteasome-ATP pathway. Several studies have shown the activation of these proteolytic pathways in cancer cachexia . Among these proteolytic pathways, the ubiquitin-proteasome-ATP-dependent pathway appears to be the most involved in cancer cachexia .This proteolytic pathway is mediated by 2 ubiquitin ligases specific for skeletal muscle, MAF-Box and MURF1, which are largely overexpressed in many models of muscular atrophy and cancer cachexia . On the other hand, the growth factor IGF1 is a known anabolic factor which activates the proteosynthesis via the signaling pathway PI3K / Akt / mTOR . The decrease in IGF1 expression in skeletal muscle is observed in experimental models of cancer cachexia . Studies have shown that certain factors of tumor origin may contribute to cancer cachexia in some animal models.

2 factors have particularly attracted the attention of scientists in recent years, the ZAG factor (Zinc alpha 2 glycoprotein), a veritable lipid mobilization factor in humans , overexpressed in the liver and adipose tissue and PIF (proteoglycan identified in mouse murine adenocarcinoma tumor cells which would be responsible for muscle wasting induced by the activation of the ubiquitin-proteasome-ATP-dependent proteolytic pathway . More recent work suggests that Myostatin and Activin A, two members of the TGFβ superfamily, may contribute to cachexia, particularly muscular atrophy, induced by certain cancers.

Adipose loss is an early syndrome in the development of cancer cachexia and is negatively correlated with patient life expectancy . Early studies on this adipose melt revealed a lack of storage of triglycerides in adipose tissue . The storage of triglycerides is achieved by the action of lipoprotein lipase. It predominantly exists in adipose tissue and hydrolyzes lipoproteins circulating in the blood, thus allowing the capture of fatty acids by adipocytes and storage of adipose reserves . The development of the tumor would induce a decrease in the gene expression and activity of lipoprotein lipase via the action of inflammatory cytokines . However, current research seems to demonstrate that the adipose melt observed in cancer cachexia is mostly explained by an increase in lipolysis (shown indirectly by an increase in plasma fatty acid concentration in cachectic patients with gastrointestinal cancer). .

Lipolysis, via hormone-sensitive lipase (LHS) and monoglyceride lipase (MGL), allows the hydrolysis of triglycerides into diglycerides and diglycerides into monoglycerides themselves degraded into free fatty acids and glycerol. Adipose tissue-specific triglyceride lipase (TGLA) has recently been discovered and has a role that is redundant to that of LHS. Studies of Cao et al. showed that the activation of LHS by catecholamines could constitute a mechanism of regulation of lipolysis during cancer cachexia. . An alteration of TGLA and LHS would also be responsible for an accumulation of DAG and TAG in the muscle of cancerous mice . A recent study showed that the invalidation of TGLA and LHS in 2 models of cachexia induced by injection of Lewis pulmonary carcinoma cells or B16 melanoma cells induced resistance to the development of cachexia by limiting adipose and muscular loss . Systemic inflammation developed during cancerous cachexia could also induce an increase in insulin resistance via TNFalpha . TNFalpha could inhibit the expression of perilipin A, a protein expressed on the surface of adipocyte lipid droplets , which plays a major role in the integrity of adipose tissue since it limits the access of enzymes involved in lipolysis to the lipid droplet . A decrease in the expression of perilipin A would induce an increase in lipolysis. In addition, a study by Stephens et al. in 2011 concluded that the number and size of intramuscular lipid droplets are increased in the presence of cancer and also increase with weight loss / adipose fat loss in other body compartments .

Myosteatosis, a pathological fatty deposit in skeletal muscle, is another characteristic of body composition, in addition to low muscle mass, which is associated with the poor prognosis of the cancer disease, in particular a decrease in overall survival and it has recently been shown that the muscle of cancer patients contains all the more adipose tissue that severe weight loss . Several studies have shown that myosteatosis is associated with an increase in insulin resistance and therefore a decrease in proteolysis via the inhibition of insulin transport of amino acids. The fat content of the muscle may be indirectly and non-invasively studied on the basis that the adipose tissue typically attenuates the radiation applied thereto. . The value of the attenuation measurements are determined by the rate at which the radiation passes through the tissue and is expressed in Hounsfield units (HU). Muscle and adipose tissue attenuation values were defined between -190 and -30 HU .

The weakening of the radiation in the muscle was correlated well with the fat content of the muscles. . Thus, the HU values defined by the CT scan may reflect the degree of intramuscular adipose tissue and are used to categorize the muscle of normal or exposed to myosteatosis . Low muscle mass and weakening of the radiation in muslce testify of high degree of myostaatosis and were identified as an independent prognostic factor for overall survival and mortality in cancer patients, respectively. . The comparison of muscle metabolism in obese and normoponded subjects showed an abolition of protein synthesis in response to insulin especially in muscle mitochondria in overweight subjects. Interestingly, muscle protein renewal was inversely correlated with fat mass. Such an observation raises the question of the possibility of a deleterious effect of fat mass on protein synthesis. The hypothesis of this lipotoxicity was confirmed by a work carried out in the rat which showed that the synthesis of the muscle proteins is slowed down when there is infiltration of fat into the muscle

At the cellular level, metabolism is governed by the mitochondria which provides 90% of our energy in the form of ATP. This energy is synthesized within oxidative phosphorylation, which consists of 2 entities (the respiratory chain and ATP synthase) and which allows the conversion, in water and ATP, of the reduced equivalents resulting from dehydrogenation reactions (and Decarboxylation) of energetic nutrients, in the presence of dioxygen (O2) and ADP, according to chemosmotic coupling theory . The decoupling of oxidative phosphorylation may be involved in involuntary weight loss. The work of Romestaing et al. Showed that weight loss following the development of a steatosis was associated with a decrease in the ATP / O2 ratio . Mitochondrial dysfunctions could therefore have a direct effect on the protein degradation observed during cancer cachexia. In addition, systemic inflammation caused by the development of the tumor can also affect mitochondrial bioenergetics.

The works of Hochwald et al. were among the first to suggest an alteration of muscle mitochondrial metabolism by demonstrating a decrease in ATP concentration in the gastrocnemius of rats with MCA sarcoma . The recent works of Constantinou and col. confirmed this hypothesis by demonstrating in vivo by 31P nuclear magnetic resonance (NMR) a reduction in the rate of synthesis of ATP on the lower limb of mice with Lewis pulmonary carcinoma compared to its healthy mice . This work suggested a decrease in the ability to synthesize ATP during cancerous cachexia through decoupling proteins such as UCP3 . This decrease in ATP synthesis could also be explained by alterations in the functioning of the mitochondrial respiratory chain .

Julienne and col. in 2012 studied the mitochondrial activity of skeletal muscles in murine models of cancer cachexia based on the ATP / Oxygen ratio and concluded that muscular mitochondrial oxidative capacities were reduced by decreasing the activity of complex IV, responsible for muscle loss and accumulation of free fatty acids in muscle (myosteatosis) since less oxidized by mitochondria. They also observed that the expression of MURF1 and MAF-Box (proteolytically active ligases) was increased in the muscle of rats with cancers .

Cancerous cachexia affects about 80% of patients with advanced cancer and increases their prognosis by increasing their morbidity and mortality. It is defined as a loss of lean mass especially muscular resulting from an imbalance between proteolysis and proteogenesis. It has been shown that the presence of cancer in the murine model favors the development of myosteatosis, which is linked, among other things, to alteration of muscle lipases and a decrease in mitochondrial activity, the consequence of which is a decrease Of the oxidation by the latter of free fatty acids which would consequently accumulate in the muscle of mice suffering from cancer. It is known that this myosteatosis then induced is responsible for an insulin resistance participating in a decrease in proteogenesis and therefore in weight loss.

The main objective here is to confirm this same hypothesis in humans by studying the influence of cachexia on muscle mitochondrial activity as a marker of myosteatosis in patients with cancer of the upper air-digestive tract, cachectic or not, and non-cachectic controls.

Patients will be recruited from ENT and Cervico-facial Surgery at CHU Gabriel Montpied in Clermont-Ferrand.

Inclusion of patients in 2 groups:

* Group K +: cancer of the upper aerodigestive tract with or without cachexia
* Group K-: absence of cancer and absence of cachexia The recruitment arrangements for the K + group will be made through a Multidisciplinary Consultation Meeting (RCP), the decision of which is an exclusive or non-exclusive surgery. Before the protocol is realized, during the preoperative consultation, an information sheet is given to the patient and an informed consent in 2 copies is signed after a period of reflection of the patient of 7 days.

At inclusion, the day before the surgery, patients benefit from a dual general and nutritional evaluation:

* Collection of epidemiological data: age, medical and surgical history (cardiac insufficiency, renal insufficiency, respiratory insufficiency, COPD, coronary artery disease), ethyl intoxication (gram / day), tobacco poisoning (package / year), usual treatment, tumor characteristics for group K+ (histological type, location, tumor stage, nature of treatment), indication and nature of surgery for group K-, pre-operative renutrition program for K + group (food supplements, enteral or parenteral feeding )
* Clinical nutritional evaluation: bodyweight (kg), weight loss in the last 6 months (kg), height (m), body mass index (BMI in kg / m²) (NPH), Short Physical Performance Battery (SPPB), muscle strength measurement by dynamometry (Newton), Impedancemetry (Kyle index, Janssen index)
* Myostéatosic and nutritional morphological evaluation by, respectively, Hounsfield Unit and Muscular Mass Index at L3 level (cm² / m²) by abdominal tomodensitometry for the K + group (carried out in the cancer extension imaging balance)

Patients will benefit from 4 organic samples during the planned surgery (carcinological surgery for Group K +, cervical surgery for Group K-):

* Carrying out a muscle biopsy of the SCOM muscle with a total volume of about 300 mg, without resorting to an additional invasive act. This sampling is immediately divided into 6 samples and placed in a liquid nitrogen tank for transport to the place of storage. It will then be frozen at -80 ° C.
* Carrying out a blood sample according to the following conditions: 1 dry tube, 1 EDTA tube and 2 dry tubes for biochemistry The dry tube and the EDTA tube will be immediately put in ice for transport to the storage site. It will then be immediately centrifuged and then frozen at -80 ° C. The two dry tubes for biochemistry will be transmitted to the laboratory of biochemistry of the CHU Gabriel-Montpied.
* Carrying out a tumor biopsy with a total volume of approximately 200 mg without resorting to an additional invasive procedure. This sampling is immediately divided into 4 samples and placed in a liquid nitrogen tank for transport to the place of storage. It is then frozen at -80 ° C (only for K + Group).

ELIGIBILITY:
Inclusion Criteria:

* For the Cancer Group (K + Group):
* Active cancer of the upper aerodigestive tract
* Eligible for surgery treatment decided by CPR
* Age ≥ 18 years or Age ≤ 80 years

For the control Group (K- Group):

* No active cancer or a history of cancer less than 5 years old - Head and neck surgery for any reason except cancer
* Absence of cachexia, defined by a weight loss> 5% over the last 6 months
* Age ≥ 18 years or Age ≤ 80 years

Exclusion Criteria:

* For groups K + and K-:
* Presence of another obvious etiology of undernutrition
* A history of heart failure, respiratory failure (requiring long-term oxygen therapy) or chronic renal disease (MDRD clearance <60 ml / min), moderate, severe or very severe COPD (HAS classification), insulin-dependent diabetes , Coronary artery disease
* Age <18 years or Age >80 years
* Protected persons and pregnant and / or nursing women

For the group K-:

- Posterior diagnosis of cancer in the case of anatomo-pathological analysis (eg thyroidectomy, parotidectomy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cancer of the upper aerodigestive tract
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
ATP / Oxygen ratio | at day 1
  The ratio of ATP produced by mitochondria and oxygen consumed by muscle mitochondria

SECONDARY OUTCOMES:
Study of enzymatic mitochondrial activity | at day 1
  (Expression of cytochrome c oxidase, citrate synthase, HAD, complexes 1, 2 and 3 of the mitochondrial respiratory chain)
Study of the activity of muscle lipases | at day 1
  (Expression of ATGL and HSL)
Study of the mobilization of the muscular lipid droplets | at day 1
  (Expression of the Perilipines 3 and 5)
Study of the muscular lipid infiltration | at day 1
  (Muscular ceramide concentration, DAG and TAG)
Study of myosteatosis | at day 1
  myosteatosis (Computed tomography in L3 for quantification in Hounsfield units)
Study of the activity of signaling pathways of protein anabolism | at day 1
  (phosphorylation rate of mTOR and EiF2alpha)
Study of the activity of the signaling pathway of insulin in the muscle | at day 1
  (AkT phosphorylation rate)
Study of muscle proteolytic activity | at day 1
  (Expression of MURF1 and MAF-box ligases)
Evaluation of the preoperative metabolic and nutritional plasma status of patients | at day 1
  (Insulinemia, Fasting Glycemia, Hepatic and Lipid Assessment, CRP, Albumin, Pre-albumin, Blood Ionogram, Inflammatory Markers)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane WALRAND, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France